CLINICAL TRIAL: NCT06475105
Title: Effects of Combination Oral Acetazolamide and Intravenous Furosemide on Acute Decompensated Heart Failure
Brief Title: Combination Oral Acetazolamide and Intravenous Furosemide on Acute Decompensated Heart Failure Outcomes
Acronym: COAF-HF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Ilham Uddin, MD, MD, FAsCC, FSCAI, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No16129/EC/KEPK-RSDK/2024
Record Dates: First submitted 2024-06-19; First posted 2024-06-26 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Oral Acetazolamide; Acute Decompensated Heart Failure; Congestion
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: This research is an experimental clinical study with a double blinded randomized controlled trial design. The study group consisted of patients with acute decompensated heart failure with volume overload who required intravenous diuretic therapy. The first group was patients who received intravenous furosemide plus acetazolamide 250 mg / 12 hours orally for up to 3 days (group A). Meanwhile, the second group was patients who received intravenous furosemide plus placebo for up to 3 days (group B).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Oral Acetazolamide) (Experimental): Participants who received intravenous furosemide plus acetazolamide 250 mg / 12 hours orally for up to 3 days.
  Interventions: Drug: Oral Acetazolamide
- Group B (Placebo) (Placebo Comparator): Participants who received intravenous furosemide plus Placebo / 12 hours orally for up to 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Acetazolamide — Participants will be randomized into group receiving either oral acetazolamide or placebo for up to 3 days
  Other Names: Glauseta
  Arms: Group A (Oral Acetazolamide)
Drug: Placebo — Participants will be randomized into group receiving either oral acetazolamide or placebo for up to 3 days
  Arms: Group B (Placebo)

SUMMARY:
Based on ADVOR trial, the potential of adding acetazolamide in increasing the success of decongestion, the amount of natriuresis and diuresis. However, the use of intravenous acetazolamide may not be possible in Indonesia, where the intravenous formulation is not available. This clinical research study is being conducted in single hospitals in Indonesia. We aim to learn if Oral Acetazolamide in addition to Furosemide intravenous works to treat congestion in Acute Decompensated Heart Failure, besides evaluating the total urinary output, change of NT pro BNP level, and safety profile of oral Acetazolamide.

The hypothesis of this study is oral acetazolamide works well to achieve successful decongestion.

DETAILED DESCRIPTION:
This is a randomized, double blind study with 2 treatment groups. Participants diagnosed with ADHF who meet the inclusion criteria and no exclusion criteria are given an explanation regarding the research and additional therapy that will be given, then informed consent is requested. Participants will be randomized to one of the two treatment groups by chance. Patients randomized to the first group will receive intravenous furosemide and oral acetazolamide. Patients randomized to the other treatment group will receive a combination of iv furosemide and placebo. It is expected that the patients of the treatment group with the combination therapy will have a faster reduction of their fluid overload. In consequence the treatment duration and total dose of diuretics administered will be shorter.

ELIGIBILITY:
Inclusion Criteria:

* Agree to be included in the research by signing informed consent
* Patients with a clinical diagnosis of acute decompensated heart failure with at least one clinical sign of volume overload with a congestion score ≥2 (ADVOR Score) (e.g. edema (score 2 or more), ascites confirmed by physical examination or ultrasonography or pleural effusion confirmed by chest x-ray or echocardiography).
* Patients on routine oral loop diuretic therapy with a dose of ≥40 mg furosemide for ≥1 month
* Plasma NT-proBNP levels that increase ≥300 pg/mL or the applicable cut-off according to the age range at the time of examination in the ER.

Exclusion Criteria:

* Subjects with acute coronary syndrome
* History of congenital heart disease requiring surgical correction.
* Subjects in cardiogenic shock.
* Estimated glomerular filtration rate <20 mL/min/1.73m² at the time of examination.
* Use of renal replacement therapy or ultrafiltration at any time before the study was included.
* Treatment with acetazolamide within 1 month before randomization.
* Exposure to nephrotoxic agents (i.e. contrast dye) is anticipated within the next 3 days
* Subjects who are pregnant or breastfeeding.
* Subjects with urinary incontinence who are unwilling to use a bladder catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful Decongestion | within 3 days
  Conditions without volume overload, no signs of excess volume within 3 days of treatment. Congestion was assessed using the volume assessment score (also called congestion score) from the ADVOR trial. The absence of fluid volume excess was defined as no more than mild edema, no residual pleural effusion, and no residual ascites. Total score ≤1 indicates that decongestion has been achieved, score >1 is considered to indicate persistent fluid volume excess (decongestion not achieved).

SECONDARY OUTCOMES:
NT pro BNP | within 3 days
  the effect of adding combination oral acetazolamide on NT pro BNP levels in ADHF participants who received iv furosemide
Renal Function | From date of randomization until the date of first documented worsening renal function (increased of creatinine serum level >50% of baseline creatinine) or date of death from any cause, evaluation every 48 hours or whichever came first, up to 90 days
  Kidney function is measured based on estimated GFR (eGFR) according to the CKD-EPI formula which is shown in units of mL/min/1.73 m2 taken on day 0, day 2, and day 4, every 48 hours during hospitalization (after receiving treatment).
Urinary Output | From date of randomization until participants discharge from hospital up to 7 days post discharge.
  the amount of urine for 24 hours is measured from the time the patient arrives at the emergency room, a urinary catheter tube is installed, measured every 24 hours during hospital treatment.
Length of Stay | From date of randomization until the date of first documented progression and discharge from hospital or date of death from any cause, whichever came first, assessed up to 30 days.
  Defined as the duration of the patient receiving treatment in hospital from the time admitted to the ER until the patient was discharged/discharged from the hospital, obtained as the date of discharge from the hospital minus the sampling date +1.

CONTACTS AND LOCATIONS:
Overall Officials: Ilham Uddin, MD, Principal Investigator — Department Cardiology and Vascular Medicine Universitas Diponegoro Kariadi General Hospital
Locations (2):
- Indonesia (2):
  - Department of Cardiology and Vascular Medicine, Universitas Diponegoro, Kariadi Central General Hospital, Semarang, Central Java
  - Kariadi Central General Hospital, Semarang, Central Java

IPD SHARING:
Plan to Share IPD: No
Currently, the decision regarding which Individual Participant Data (IPD) will be included for sharing is still under consideration. This undecided status is due to several key factors that require thorough evaluation